CLINICAL TRIAL: NCT00885794
Title: Microperimetry and High-Definition-OCT in Ranibizumab Treatment for Diabetic Macular Edema (MORE-Study)
Brief Title: Microperimetry and Optical Coherence Tomography (OCT) With Lucentis for Diabetic Macular Edema (DME)
Acronym: MORE
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery (Other)
Responsible Party: Priv. Doz. OA Dr. Ulrike Stolba, Department of Ophthalmology, The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery, Rudolf Foundation Clinic
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: EK 08-069-0508
Record Dates: First submitted 2009-04-20; First posted 2009-04-22 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Diabetic Macular Edema
Keywords: Clinically Significant Diabetic Macular Edema; Focal Laser; GRID-Laser; Ranibizumab; Lucentis; Microperimetry; High-Definition OCT; Randomized; Observer-Blinded; Ineffective Treatment with Focal Laser or GRID-Laser
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.5 mg Ranibizumab (Experimental): 3 intravitreal injections of 0.5 mg Ranibizumab every 5 weeks
  Interventions: Drug: Ranibizumab
- 1.0 mg of Ranibizumab (Experimental): 3 intravitreal injections of 1.0mg Ranibizumab every 5 weeks
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — 3 intravitreal injection every 5 weeks
  Other Names: Lucentis

SUMMARY:
Diabetic maculopathy is the leading cause of visual impairment in the working-age population in developed countries. Diabetic macular edema can cause impaired visual acuity and so far is treated by laser, vitreous surgery, and intravitreal cortisone application. Still 50% of the cases do not respond to the treatment.

Recently intraocular anti-VEGF-treatment with ranibizumab (Lucentis®, Novartis) in diabetic macular edema has proven efficacy to last over a period of 3 to 6 months. Still, the optimal dosage for those intravitreal injections still has to be found, because frequent injections are necessary.

The measurement of visual acuity is inadequate to quantify in detail the visual impairment. Using the newest technology of a high-definition optical coherence tomography (Cirrus-OCT, Carl Zeiss Meditec Inc.) to determine the retinal thickness, and a miroperimetry (MP-1, Nidek Technologies) to determine retinal sensitivity, we hope to find the optimal dosage of intravitreal anti-VEGF treatment in diabetic macular edema.

Study objective: To determine the dose response of 0.5mg and 1.0mg ranibizumab (Lucentis®, Novartis Pharma) intravitreal injection in subjects with resistant diabetic macular edema and evaluate safety and tolerability.

DETAILED DESCRIPTION:
Diabetic maculopathy due to diabetic macular edema (DME) is the leading cause of visual impairment in the working-age population in developed countries. DME is the swelling of the retina resulting from the exudation and accumulation of extracellular fluid and proteins in the macula. Structural changes in the endothelium of retinal vessels lead to a breakdown of the blood-retina barrier and increase vascular permeability, resulting in exudation. The standardized treatment of DME is a focal laser or GRID-laser treatment with or without combined triamcinolone intravitreal injections. Those laser treatments produce scars in the central retina and are not always very effective. In cases of macular traction or taut posterior hyloid vitrectomy and retinal surgery are necessary.

Vascular endothelial growth factor (VEGF) has been implicated as an important factor in the occurrence of vascular permeability in DME. In patients with DME, VEGF levels are significantly elevated, compared to patients without ocular disease. Therefore, anti-VEGF treatment has been implicated as an important treatment of DME and recently intraocular anti-VEGF-treatment with ranibizumab (Lucentis®, Novartis Pharma) in diabetic macular edema has proven to be very effective. Just like in patients with age-related macular degeneration (AMD), anti-VEGF treatment was given 3 times every 4-6 weeks. The same treatment was repeated at a relapse of the disease, again 3 times every 4-6 weeks. One study group treated DME with 0.5mg ranibizumab intravitreal injections and the other compared 0.3mg to 0.5mg of ranibizumab intravitreal injections. An optimal treatment dose has not been found yet.

Visual acuity assessment is currently used to determine the functional damage caused by edema, although it may not completely describe the functional condition of the patient. Furthermore, visual acuity alone does not seem to be the best parameter to define the effect and continuation of treatment. Retinal thickness, as measured by the noninvasive optical coherence tomography (OCT) can deliver detailed information about the retinal situation during and after treatment. Also a fundus related perimetry, known as microperimetry (MP), is a useful noninvasive examination method in determining the site of relative and absolute scotomas and also fixation characteristics. With MP the macular sensitivity can be measured to further assess the macular condition.

Using the newest technology of a high-definition OCT (Cirrus-OCT, Carl Zeiss Meditec Inc.) to determine the retinal thickness, and a MP with automated correction for eye movements (MP-1, Nidek Technologies) to determine retinal sensitivity, we intend to analyze this new treatment option for DME, and find the optimized dose for intravitreal injection of ranibizumab in cases of ineffective laser treatment.

ELIGIBILITY:
Inclusion Criteria:

* Study eye with clinically significant macular edema, for which one of the following characteristics has to be present:
* retinal thickening at or within 500µm from the center of the macula,
* hard exudates at or within 500µm from the center of the macula associated with thickening of the adjacent retina,
* a zone (>1-disk area) or zones of retinal thickening of which any part is within 1 disk diameter from the center of the macula.
* Second line treatment after ineffective laser treatment
* Men or women with diabetes mellitus
* Only one eye per patient
* Age > 50 years
* HbA1c < 8%

Exclusion Criteria:

* Study eye with concomitant retinal or choroidal disorder other than diabetic retinopathy
* Study eye with significant central lens opacities and / or conditions that limit the view of the fundus
* poor general condition
* woman of childbearing potential, current pregnancy or breastfeeding
* Patients who are unwilling to adhere to visit examination schedules
* Evidence of macular traction or taut posterior hyloid.

Min Age: 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-05; Primary Completion 2011-05 (Actual); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Retinal thickness | at 3 months

SECONDARY OUTCOMES:
Retinal sensitivity | 3, 6, and 9 months
Distance best corrected visual acuity | 3, 6, and 9 months
Reading best corrected visual acuity | 3, 6, and 9 months
Intraocular pressure | 3, 6, and 9 months
Type of diabetic macular edema | 3, 6, and 9 months
Type of diabetes mellitus HbA1c | 3, 6, and 9 months
Blood-pressure | 3, 6, and 9 months
Age | 3, 6, and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Stolba, MD, Principal Investigator — Department of Ophthalmology, Ludwig Boltzmann Institute for Retinology and Biomicroscopic Lasersurgery, Rudolf Foundation Clinic
Locations (1):
- Rudolf Foundation Clinic, Vienna, Vienna, Austria